CLINICAL TRIAL: NCT07340463
Title: The Efficacy and Safety of Biologics (Belimumab/ Telitacicept) Induction Therapy in Proliferative Lupus Nephritis Patients for 6 Months Compared With Mycophenolate Mofetil Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Professor, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024LCYXXH009
Record Dates: First submitted 2025-12-25; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE); Lupus Nephritis (LN)
Keywords: SLE; LN; Belimumab; Lupus Nephritis; Telitacicept
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Glucocorticoids; Adrenal Cortex Hormones; belimumab; telitacicept; Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biologics Group (Experimental): Glucocorticoids combined with a biologic agent (Belimumab or Telitacicept). All subjects receive oral glucocorticoids (starting dose 0.5 mg/kg/day, ≤40 mg/day, planned taper to ≤5 mg/day by Month 4). Combined with one biologic agent: Belimumab (IV infusion, 10 mg/kg/dose, every 2 weeks) or Telitacicept (subcutaneous injection, 160 mg/dose, once weekly). The specific biologic is chosen through discussion between the investigator and the patient. If no response after 3 months of induction therapy, subjects may switch to the Triple Therapy Group.
  Interventions: Drug: Glucocorticoids; Biological: belimumab; Biological: Telitacicept
- Standard of Care (SOC) Group (Active Comparator): Glucocorticoids combined with Mycophenolate Mofetil (Standard of Care regimen). All subjects receive the same oral glucocorticoid regimen as the Biologics Group. Combined with Mycophenolate Mofetil (MMF), target dose 1.5-2.0 g/day, administered orally in two divided doses. If no response after 3 months of induction therapy, subjects may switch to the Triple Therapy Group.
  Interventions: Drug: Glucocorticoids; Drug: Mycophenolate mofetil (MMF)
- Triple Therapy Group (Experimental): Glucocorticoids combined with Mycophenolate Mofetil and a biologic agent (Belimumab or Telitacicept). All subjects receive the same oral glucocorticoid regimen as the other groups. Combined with Mycophenolate Mofetil (MMF) (target dose 1.5-2.0 g/day) and one biologic agent (Belimumab, every 2 weeks; or Telitacicept, once weekly). The specific biologic is chosen through discussion between the investigator and the patient. This group is both one of the initially randomized arms and the rescue therapy arm for non-responders from the other two groups.
  Interventions: Drug: Glucocorticoids; Biological: belimumab; Biological: Telitacicept; Drug: Mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: Glucocorticoids — Background therapy for all study arms. All subjects receive glucocorticoid therapy. The oral starting dose is prednisone 0.5 mg/kg/day (or equivalent), not exceeding 40 mg/day. Planned taper to ≤5 mg/day by Month 4, with stable dosing from Months 5-6. The tapering speed is determined by investigator assessment during the study. Permitted at investigator's discretion: intravenous methylprednisolone pulse therapy (dose 0.25-3.0g).
  Other Names: Corticosteroids
Biological: belimumab — A humanized monoclonal antibody targeting B-cell activating factor (BAFF). Used in the "Biologics Group" and the "Triple Therapy Group". Administered via intravenous infusion every 2 weeks at a dose of 10 mg/kg (600mg/dose) for 6 months. Premedication with dexamethasone and antihistamines is required for the first infusion to prevent allergic reactions (dexamethasone may be omitted for subsequent infusions if no prior reaction).
  Other Names: Benlysta
  Arms: Biologics Group; Triple Therapy Group
Biological: Telitacicept — A TACI-Fc fusion protein that neutralizes both BAFF and APRIL cytokines. Used in the "Biologics Group" and the "Triple Therapy Group". Administered via subcutaneous injection once weekly at a dose of 160mg for 6 months.
  Arms: Biologics Group; Triple Therapy Group
Drug: Mycophenolate mofetil (MMF) — An immunosuppressive agent. Used in the "Standard of Care (SOC) Group" and the "Triple Therapy Group". Administered orally in two divided daily doses, target dose 1.5-2.0 g/day. Maintained at the target dose until the end of the treatment period. Dose adjustment or brief interruption (preferably not exceeding 14 days) is permitted in case of specific hematologic toxicity or infectious complications.
  Arms: Standard of Care (SOC) Group; Triple Therapy Group

SUMMARY:
1. Study Design This is a single-center, prospective, randomized, controlled, exploratory clinical trial. The study is designed to evaluate and compare the efficacy and safety of two biologic-based induction regimens against standard of care (SOC) and a triple-combination regimen in patients with active proliferative lupus nephritis (LN).
2. Study Objectives Primary Objective: To compare the 6-month complete renal response (CRR) rate among patients receiving biologic-based induction therapy, SOC induction therapy, and triple-combination induction therapy.

   Secondary Objectives: To compare the rates of partial renal response (PRR) and overall renal response (ORR) at monthly intervals up to Month 6; to assess the time to achieve CRR/PRR; to evaluate changes in clinical and immunological parameters from baseline; and to compare the safety profiles of the three treatment regimens.
3. Key Eligibility Criteria Patients aged 14-65 years with biopsy-proven active Class III or IV (±V) LN according to ISN/RPS 2018 classification, an SLE-DAI score >6, and 24-hour urine protein >1.0 g/d will be eligible. Key exclusion criteria include an eGFR ≥45 ml/min/1.73m², recent use of renal replacement therapy or potent immunosuppressive procedures, significant concurrent infections, severe hematological/ hepatic abnormalities, and known hypersensitivity to the study biologics.
4. Treatment Groups and Intervention

   Eligible patients will be randomized in a 2:2:1 ratio to one of three treatment arms for a 6-month induction period:

   Biologics Group (n≈20): Glucocorticoids + either Belimumab or Telitacicept. SOC Group (n≈20): Glucocorticoids + Mycophenolate Mofetil (MMF). Triple Therapy Group (n≈10): Glucocorticoids + MMF + either Belimumab or Telitacicept.

   The choice between Belimumab and Telitacicept within the Biologics and Triple Therapy groups will be determined jointly by the investigator and the patient.
5. Study Medications & Administration Glucocorticoids: All patients will receive oral prednisone (or equivalent) starting at 0.5 mg/kg/day (max 40 mg/day), with a mandatory taper to ≤5 mg/day by Month 4 and stable dosing from Months 5-6. Intravenous methylprednisolone pulses are permitted per investigator discretion.

   Mycophenolate Mofetil (MMF): Administered only in the SOC and Triple Therapy groups. The target dose is 1.5-2.0 g/day, maintained until the end of the treatment period.

   Belimumab: Administered via intravenous infusion at 10 mg/kg (600 mg/dose) every 2 weeks.

   Telitacicept: Administered via subcutaneous injection at 160 mg once weekly. Patients in the Biologics or SOC groups showing no response by Month 3 may directly switch to the Triple Therapy regimen.
6. Primary Efficacy Endpoint

The primary endpoint is the proportion of patients achieving Complete Renal Response (CRR) at Month 6. CRR is strictly defined as:

24-hour urine protein <0.5 g/d, AND Estimated Glomerular Filtration Rate (eGFR) ≥85% of the baseline value, AND No requirement for rescue therapy or premature treatment withdrawal. 7. Secondary Efficacy & Safety Assessments Key secondary efficacy assessments include monthly CRR, PRR, and ORR rates; time to response; incidence of renal-related events; and changes in proteinuria, eGFR, serum creatinine, and disease activity scores (SELENA-SLEDAI, BILAG-2004, PGA). Safety will be evaluated through the incidence and severity of adverse events, with special attention to infections, infusion/injection reactions, and metabolic parameters.

8. Statistical Considerations This is an exploratory study with a planned enrollment of 40-50 patients. The primary analysis will use the Full Analysis Set (FAS) under the intention-to-treat principle. The difference in the Month 6 CRR rate among the three groups will be analyzed using the Chi-square test. Time-to-event data will be analyzed using the Kaplan-Meier method with Log-rank test for comparisons.

9. Hypothesis: This study protocol outlines a head-to-head comparison of novel biologic-based induction strategies against current SOC for active LN. It aims to generate critical preliminary data on whether glucocorticoids combined with a biologic (Belimumab or Telitacicept) alone can induce effective renal remission, potentially offering a targeted treatment option with a different safety profile compared to conventional immunosuppressive therapy. The results may inform the design of larger, confirmatory trials in LN management.

ELIGIBILITY:
Inclusion Criteria:

* 1.Signed written informed consent form. 2.Age 14-65 years (inclusive), any gender. 3.Meets the American College of Rheumatology (ACR) SLE diagnostic criteria (1997).

  4.All patients have biopsy-confirmed class III/IV ± V LN within the past six months.

  5.SLE-DAI score > 6. 6.Urine protein quantification > 1.0 g/d.

Exclusion Criteria:

* 1.Estimated glomerular filtration rate (eGFR) ≥45 ml/min/1.73 m². 2.Patients who have received renal replacement therapy, plasma exchange, immunoadsorption, or high-dose intravenous immunoglobulin (100g) within the past 2 months.

  3.Patients with concomitant critical organ damage or lupus crisis (e.g., pulmonary hemorrhage, encephalopathy, heart failure) deemed unsuitable for clinical trial participation by the investigator.

  4.Hematological abnormalities: White blood cells <3000/μL, absolute neutrophil count <1500/μL, or lymphocytes <800/μL, platelet count <50,000/μL (unless due to SLE activity).

  5.Liver function abnormalities: ALT, AST, or bilirubin levels exceeding 2 times the upper limit of normal.

  6.Known allergy or contraindication to any component of belimumab and/or telitacicept.

  7.Active infection or intravenous antibiotic use within 1 month prior to enrollment.

  8.Pregnant or breastfeeding women. 9.Current or within the past 3 months: Active hepatitis B, hepatitis C, tuberculosis, cytomegalovirus pneumonia, active fungal infection, syphilis infection, or HIV infection; active peptic ulcer; history of drug abuse or alcoholism; severe malnutrition (BMI <16 kg/m²).

  10.Other conditions: Severe cardiovascular disease potentially life-threatening; chronic obstructive pulmonary disease, or asthma/allergic diseases requiring long-term oral steroid treatment; malignant hypertension; history of malignancy within the past 5 years (except for completely treated basal cell or squamous cell skin cancer or cervical intraepithelial neoplasia).

  11.Other situations deemed unsuitable for enrollment by the investigator.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Complete Renal Response (CRR) Rate at Month 6 | From Baseline to Month 6
  Proportion of patients achieving Complete Renal Response. CRR is defined as: 24-hour urine protein < 0.5 g/d, AND estimated glomerular filtration rate (eGFR) ≥ 85% of the baseline value, AND no receipt of rescue therapy or premature withdrawal from treatment.

SECONDARY OUTCOMES:
Partial Renal Response (PRR) Rate at Months 1, 2, 3, 4, 5, and 6 | From Baseline to Months 1, 2, 3, 4, 5, and 6
  Proportion of patients achieving Partial Renal Response. PRR is defined as: ≥50% reduction in 24-hour urine protein from baseline, AND eGFR ≥ 85% of the baseline value, AND no receipt of rescue therapy or premature withdrawal from treatment.
Overall Renal Response (ORR) Rate at Months 1, 2, 3, 4, 5, and 6 | From Baseline to Months 1, 2, 3, 4, 5, and 6
  Proportion of patients achieving Overall Renal Response. ORR is defined as achieving either Partial Renal Response (PRR) or Complete Renal Response (CRR).
Time to Achieve Complete or Partial Renal Response | From randomization up to Month 6
  Time from randomization to the first achievement of either Complete Renal Response or Partial Renal Response.
Proportion of Patients with Renal-Related Events by Month 6 | From Baseline to Month 6
  Proportion of patients experiencing at least one renal-related event. Renal-related event is defined as: ① Death; ② Worsening proteinuria (≥50% increase in 24-hour urine protein from baseline AND value ≥3 g/g); ③ Worsening eGFR (≥30% decrease in eGFR from baseline AND value <60 mL/min/1.73 m²); ④ Receipt of rescue therapy.
Change from Baseline in 24-hour Urine Protein Quantification | Baseline, Months 1, 2, 3, 4, 5, and 6
  Absolute change and ratio from baseline in 24-hour urine protein (g/d) at each visit.
Change from Baseline in Estimated Glomerular Filtration Rate | Baseline, Months 1, 2, 3, 4, 5, and 6
  Change from baseline in estimated glomerular filtration rate (eGFR, mL/min/1.73 m²) at each visit.
Incidence of Adverse Events During the Treatment Period | From first dose until 30 days after the last dose or the Month 6 visit, whichever is later
  Proportion of patients experiencing at least one adverse event, serious adverse event, or adverse event of special interest (e.g., infusion/injection reactions, infections, new-onset hypertension/diabetes). Assessed based on abnormal findings in physical exams, vital signs, and laboratory tests (complete blood count, biochemistry, urinalysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Ethics Committee of the General Hospital of Eastern Theater Command of the People's Liberation Army, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided